CLINICAL TRIAL: NCT00464373
Title: Injection of Botulinum Toxin Type A Into the External Urethral Sphincter for Male Patients Suffering From Chronic Prostatitis/Chronic Pelvic Pain Syndrome (NIH Cat. III): a Prospective, Double-blind and Placebo-controlled Clinical Trial
Brief Title: Botulinum Toxin Type A for the Treatment of Male Chronic Pelvic Pain Syndrome
Acronym: BTX-URO-01
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow accrual.
Sponsor: Daniel Stephan Engeler (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor-Investigator, Daniel Stephan Engeler, Dr. med., Cantonal Hospital of St. Gallen
Organization: Cantonal Hospital of St. Gallen (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BTX-URO-01; EKSG 06/056
Record Dates: First submitted 2007-04-20; First posted 2007-04-23 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2014-01

CONDITIONS: Chronic Prostatitis With Chronic Pelvic Pain Syndrome; Prostatitis
Keywords: Prostatitis; Chronic Prostatitis with Chronic Pelvic Pain Syndrome; Botulinum Toxin Type A; Drug therapy; Injections, intramuscular
MeSH Terms: conditions — Prostatitis | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Botulinum Toxin Type A 200 U in 4ml NaCl 0.9%
  Interventions: Drug: Botulinum Toxin Type A
- 2 (Placebo Comparator): 4ml NaCl 0.9%
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Botulinum Toxin Type A — Single intrasphincteric injection at the 3,6,9, and 12 o'clock positions of the external urethral sphincter (1 ml of drug solution each)
  Other Names: Botox
  Arms: 1
Drug: Placebo — 4ml NaCl 0.9%
  Arms: 2

SUMMARY:
The aim of this randomized placebo-controlled study is to demonstrate the efficiency and safety of the injection of Botulinum Toxin Type A (200 Units) into the external urethral sphincter for the treatment of chronic prostatitis/chronic pelvic pain.

DETAILED DESCRIPTION:
The treatment of the male CP/CPPS is often as unsuccessful as frustrating for patients and doctors. Because of that patients change their general practitioners or urologists quite regularly. One of the major problems is the unknown pathomechanism of the disease. Most patients are suffering from irritative voiding symptoms and a dysfunction of the pelvic floor. By looking at the various (non-) conservative therapeutical strategies it becomes quite clear that there is no unique and convincing therapeutical strategy.

At present Botulinum-Toxin Type A (BTX A) is widely used in the urological field especially for para-/tetraplegics patients having trouble with neurogenic bladder dysfunction. It has been reported in case series (doses: 200U and 30U) that BTX A injected into the external urethral sphincter is able to reduce the symptoms without provoking incontinence. This is implied with the hypothesis that obstructive voiding symptoms because of a CP/CPPS are associated with an incomplete relaxation of the bladder neck and the external urethral sphincter.

After having given their informed consent, patients undergo a screening visit and baseline evaluation including patients history, clinical examination, NIH-CPSI and IPSS-questionnaires, micturition diary, sonography, 4-glass test and urodynamics. Patients fulfilling the study eligibility criteria are randomized to receive intrasphincteric injection of either BTX A or placebo. There will be 5 follow-up visits including a post-treatment follow-up after 1 year.

ELIGIBILITY:
Inclusion Criteria:

* CPPS NIH III (symptoms over 3 months during the last 6 months, 4 glass-test)
* Pain Score ≥ 4

Exclusion Criteria:

* During the last month: intake of antibiotics, alpha receptor blockers, anticholinergics; intake of analgesics containing opioids (longer than 4 days); participating in a different clinical trial
* During the last 3 months:documented urinary infection, epididymitis, positive urinary culture; status post biopsy of the prostate gland; STD: Gonorrhea, Chlamydia, Mycoplasm, Trichomonads
* During the last 6 months: Finasteride or any other 5α-reductase inhibitor
* During the last 12 months: status post any surgery on the prostate gland; genital herpes; not adjustable hypertension, angina pectoris, heart failure (NYHA III-IV), Status post myocardial infarction, coronary bypass surgery or coronary dilatation
* During the last 24 months: cerebral insult, TIA; active disease of the liver
* Other urological diseases like prostate cancer, bladder cancer, status post radiation of the small pelvis, chemotherapy (intravesical or systemic)
* Urinary catheter
* Residual urine > 200ml
* Serum creatinine > 200µmol/l
* Status post injection of BTX A, hypersensitivity concerning any substances of content of BTX, myasthenia gravis
* Any kind of cancer
* Active inflammation (except the prostate gland)
* Neurological or psychological disease making signing of a consent form or behaving according to a study protocol impossible
* Abuse of drugs or alcohol during last 5 years
* Any disease that may influence the results according to the opinion of the medical doctor

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2007-04; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
NIH-CPSI Total Score | 1 year

SECONDARY OUTCOMES:
NIH-CPSI Subscales | 1 year
Standardized questions for the assessment of the treatment outcome | 1 year
International prostate symptom score (I-PSS) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S Engeler, MD, Principal Investigator — Department of Urology, Cantonal Hospital of St. Gallen, St. Gallen, Switzerland; Hans-Peter Schmid, MD, Study Director — Department of Urology, Cantonal Hospital of St. Gallen
Locations (1):
- Department of Urology, Cantonal Hospital of St. Gallen, Sankt Gallen, Canton of St. Gallen, Switzerland